CLINICAL TRIAL: NCT03908411
Title: The Effect of Paratracheal Pressure on the Glottic View During Direct Laryngoscopy : a Randomized Controlled Trial
Brief Title: The Effect of Paratracheal Pressure on the Glottic View
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 10-2019-16
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Paratracheal Pressure; Sellick's Maneuver; Airway Management; Cricoid Pressure
Keywords: Paratracheal pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paratracheal pressure (Active Comparator): Left Paratracheal pressure is applied by ultrasound transducer after confirmation of the location of the esophagus.
  Interventions: Procedure: Paratracheal pressure
- Sellick's maneuver (Active Comparator): Conventional Sellick's maneuver is applied.
  Interventions: Procedure: Sellick's maneuver

INTERVENTIONS:
Procedure: Paratracheal pressure — Paratracheal pressure is applied by 30N force with the ultrasound transducer.
  Arms: Paratracheal pressure
Procedure: Sellick's maneuver — Conventional Sellick's maneuver is applied by 30N force
  Arms: Sellick's maneuver

SUMMARY:
Paratracheal pressure may have a role in the prevention of pulmonary aspiration. The effects of paratracheal pressure on glottic view, ease of facemask ventilation, or tracheal intubation are not studied yet. In this study, the subjects are divided into two groups (group I: paratracheal pressure applied during induction of anesthesia, group II: conventional Sellick's maneuver applied during induction of anesthesia). Investigators will assess the glottic view during direct laryngoscopy.

DETAILED DESCRIPTION:
Primary outcome:

-Cormack-Lehane grade

Secondary outcome:

* POGO score before and after application of each intervention
* Difficulties of mask ventilation after application of each intervention
* Inspiratory pressure and tidal volume during manual mask ventilation
* Rates of worsening of the glottic view after intervention
* The difficulty of endotracheal intubation
* Intubation time

ELIGIBILITY:
Inclusion Criteria:

Adult patient undergoing elective surgery with general anesthesia

Exclusion Criteria:

A patient who does not agree to participate in this study A patient who has a history of cervical/esophageal operation A patient who has a risk of gastric regurgitation A patient who has atherosclerosis of the left carotid artery or history of stroke or angina in 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Cormack-Lehane grade | During anesthesia induction procedure
  Cormack-Lehane grade

SECONDARY OUTCOMES:
POGO | During anesthesia induction procedure
  The percentage of glottic opening (POGO), linear span from the anterior commissure to the interarytenoid notch, 0-100%, higher value represent a better view
Difficulty of mask ventilation | During anesthesia induction procedure
  Difficulty of mask ventilation evaluated by the anesthesiologist (Easy/Moderate/Difficult/Impossible)
Inspiration pressure | During anesthesia induction procedure
  Pressure to maintain adequated ventilation after application of the intervention
Tidal volume | During anesthesia induction procedure
  Tidal volume which is achieved after application of the intervention
Intubation difficulty | During anesthesia induction procedure
  Subjective evaluation of the difficulty to pass the endotracheal tube into the glottic opening, easy/moderate/difficult

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - SMG - SNU Boramae Medical Center, Seoul

REFERENCES:
- [Derived] Won D, Kim H, Chang JE, Lee JM, Min SW, Ma S, Kim C, Hwang JY, Kim TK. Effect of Paratracheal Pressure on the Glottic View During Direct Laryngoscopy: A Randomized Double-Blind, Noninferiority Trial. Anesth Analg. 2021 Aug 1;133(2):491-499. doi: 10.1213/ANE.0000000000005620. PMID 34081034